CLINICAL TRIAL: NCT02654522
Title: The Use of a Recombinant DNA-based Hyaluronidase (RDNAH/ Hylenex Recombinant) to Dissolve Fixed Amounts of a Variety of Popular Hyaluronic Acid (HA) Dermal Fillers in Human Subjects.
Brief Title: The Use of a Recombinant DNA-based Hyaluronidase to Dissolve Fixed Amounts of Hyaluronic Acid Dermal Fillers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Steve Yoelin M.D. Medical Associates, Inc. (Other)
Responsible Party: Principal Investigator, Steven Yoelin, Steve Yoelin M.D., Steve Yoelin M.D. Medical Associates, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HH101
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Dermal Filler
MeSH Terms: interventions — Hyaluronoglucosaminidase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Filler (Experimental): Each subject will have one product in one forearm and another product in the other. Products: JUVEDERM Ultra Plus (24 mg/mL of HA) and VOLUMA (20 mg/mL of HA). Subjects will be randomized as to which forearm will receive which product. In one forearm, subject will receive four injections of the assigned HA filler (0.2mL). HA injections will be placed along a line from the wrist to the antecubital fossa. The initial 0.2mL HA injection will be placed in the deep dermis 5 cm from the wrist and the subsequent three 0.2mL HA injections will be place in 5 cm increments in the deep dermis along the line noted above. Same process will be used on the contralateral forearm using the other HA filler.1-3 hours post injection, these 8 HA injection sites (4 per forearm) per subject will then receive a randomized amount of Hylenex recombinant (0U, 30U, 60U or 75U).
  Interventions: Drug: Hylenex
- Scale Validation (No Intervention): One forearm of one of three subjects will be randomized to the scale "control" forearm. The opposite forearm of this subject as well as the forearms of the two remaining subjects will receive treatment in this study. The forearm that has been designated as the scale "control" forearm will be injected with VOLUMA in a straight line into the mid-dermis in the following manner: 0.05ml of VOLUMA will be injected 5 cm proximal to the wrist, 0.1ml of VOLUMA will be injected 10 cm proximal to the wrist, 0.15ml of VOLUMA will be injected 15 cm proximal to the wrist and 0.2ml of VOLUMA will be injected 20 cm proximal to the wrist. The remaining "randomized" forearms (the non-injected forearm from the subject above and the forearms from the two additional subjects) will be injected in a similar fashion to the "control" forearm as noted above; however, the dose at each location will be randomized. Control subject will receive no Hylenex until after pertinent data is collected for the study.

INTERVENTIONS:
Drug: Hylenex — 1-3 hours post injection, the 8 HA injection sites (4 per forearm) per subject will then receive a randomized amount of Hylenex recombinant (0U, 30U, 60U or 75U).
  Other Names: Hyaluronidase
  Arms: Filler

SUMMARY:
The purpose of this study is to determine whether or not Recombinant DNA-based hyaluronidase (RDNAH/Hylenex recombinant), is safe and effective for dissolving hyaluronic acid (HA) dermal fillers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Able to speak/write in the English language
* Negative Pregnancy Test on Day 1
* Proposed injection site must be free of any active inflammation

Exclusion Criteria:

* Pregnant or breast feeding
* History of keloid formation
* History of allergic reaction to hyaluronic acid dermal fillers, hyaluronidase, or any ingredients of the aforementioned products
* Active, uncontrolled inflammatory condition of any type
* History of allergic reaction to lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Cutaneous Augmentation Grading Scale (Vartanian et al, 2005) | 2-6 hours post initial injection

SECONDARY OUTCOMES:
Photography (Volar Aspect) at Site of Injection | 1-6 hours post initial injection day 1, day 2
3-dimensional (3-D) ultrasound imaging | 1-6 hours post initial injection day 1, day 2

CONTACTS AND LOCATIONS:
Overall Officials: Steven G Yoelin, M.D., Principal Investigator — Steve Yoelin M.D. Medical Associates, Inc.